CLINICAL TRIAL: NCT06506214
Title: Cross-sectional Multicenter Study Aimed at Characterizing Adherence to Treatment and Satisfaction With Care in Patients With Cutaneous Lupus
Brief Title: Characterizing Adherence to Treatment and Satisfaction With Care in Patients With Cutaneous Lupus
Acronym: ADlupus
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/22/0298
Record Dates: First submitted 2024-07-11; First posted 2024-07-17 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Cutaneous Lupus
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — Responses to questionnaires:
  * Cutaneous Lupus Erythematosus Disease Area and Severity Index (CLASI)
  * Medical Adherence Self-Report Inventory (MASRI)
  * Morisky Medication Adherence Scale (MMAS4)
  * Visual analog scale (VAS) on the perception of disease control
  * Belief on Medicine Questionnaire (BMQ)
  * Care patient Feedback measure
  * Hospital Anxiety and Depression Scale (HAD)
  * Dermatology Life Quality Index (DLQI)

SUMMARY:
This multicenter study aims to evaluate treatment adherence and satisfaction of patients with cutaneous lupus, influenced by perception of the disease, fear of side effects, cost of medications and the doctor-patient relationship. Adherence will be measured by a VAS of 80% or higher on the Medical Adherence Self-Report Inventory scale.

DETAILED DESCRIPTION:
This multicenter, cross-sectional study aims to characterize adherence to treatment and satisfaction of patients with cutaneous lupus. Non-adherence to treatment is a major problem, influenced by perception of the disease, fear of adverse effects, cost of medications and the doctor-patient relationship. Adherence will be measured by a VAS of 80% or more on the visual analog scale of the Medical Adherence Self-Report Inventory questionnaire.

The study is descriptive, multicenter and cross-sectional. Participants will be adult patients suffering from cutaneous lupus, diagnosed by a dermatologist and under treatment, able to complete questionnaires. Patients with systemic lupus, cognitive or psychiatric disorders will be excluded from the study.

The inclusion period is two years, with 30 minutes of follow-up per participant. The study will provide a better understanding of the feelings of patients with cutaneous lupus and the factors limiting their adherence to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cutaneous lupus (pure cutaneous or subacute) diagnosed by a dermatologist and under local and/or systemic treatment for cutaneous lupus
* No opposition to participation
* Patient able to complete the questionnaires
* Adult patient

Exclusion Criteria:

* Systemic lupus with multiple visceral involvement
* Cognitive or psychiatric disorders preventing the smooth running of the study
* Pregnant woman
* Patient under guardianship/curatorship or safeguard of justice

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with cutaneous lupus (pure cutaneous or subacute) diagnosed by a dermatologist and under local and/or systemic treatment for cutaneous lupus.
Sampling Method: Non-Probability Sample
Enrollment: 233 (Estimated)
Dates: Start 2022-10-08 (Actual); Primary Completion 2024-10-08 (Estimated); Study Completion 2024-10-08 (Estimated)

PRIMARY OUTCOMES:
Evaluation of adherence to treatment of patients with cutaneous lupus. | Inclusion day
  Adherence is defined by a VAS greater than or equal to 80% on the Visual Analog Scale of the MASRI (Medical Adherence Self-Report Inventory) questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Carle PAUL, MD, Principal Investigator — University Hospital, Toulouse
Locations (4):
- France (4):
  - University Hospital Montpellier, Montpellier
  - APHP Hôpital Saint-Louis, Paris
  - Hôpital Tenon, Paris
  - University Hospital Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No